CLINICAL TRIAL: NCT00449072
Title: A Randomized, Multicenter, Double-blind, Placebo-controlled, Parallel Group Study of the 12 Month Effect of Treatment With Once Daily Triamcinolone Acetonide (NASACORT® AQ Nasal Spray 110 μg) on the Growth Velocity of Children, 3 to 9 Years of Age, With Perennial Allergic Rhinitis (PAR)
Brief Title: Study of Triamcinolone Acetonide on the Growth Velocity of Children, Ages 3 to 9, With Perennial Allergic Rhinitis (PAR)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XRG5029C_3503
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Results first posted 2012-08-07 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2011-10

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Loratadine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): 3 to 9 year old participants with Perennial Allergic Rhinitis (PAR) administered
  * Placebo in the baseline/screening period to demonstrate administration of investigational product (IP) with the nasal spray bottle
  * Placebo in the double-blind treatment period
  All participants were provided Children's Claritin® Syrup as a rescue medication.
  Interventions: Other: Placebo; Drug: Claritin®
- TAA-AQ (Active Comparator): 3 to 9 year old participants with Perennial Allergic Rhinitis (PAR) administered
  * Placebo in the baseline/screening period to demonstrate administration of IP with the nasal spray bottle
  * Triamcinolone acetonide (TAA-AQ) in the double-blind treatment period
  All participants were provided Children's Claritin® Syrup as a rescue medication.
  Interventions: Other: Placebo; Drug: TAA-AQ, Nasacort® AQ; Drug: Claritin®

INTERVENTIONS:
Other: Placebo — Placebo to TAA-AQ was administered once at the study site in each nostril during the baseline/screening period to demonstrate intranasal IP administration
Other: Placebo — Placebo to TAA-AQ was administered intranasally once daily in each nostril during the double-blind period
  Arms: Placebo
Drug: TAA-AQ, Nasacort® AQ — 110 μg TAA-AQ was administered once daily intranasally (1 spray delivering 55 μg of TAA-AQ in each nostril) during the double-blind treatment period
  Arms: TAA-AQ
Drug: Claritin® — Participants were provided Children's Claritin® Syrup (5 mg of loratadine per 5 mL), as rescue medication for the relief of allergic rhinitis (AR) symptoms, and could be used throughout the study on an as needed basis according to the Food and Drug Administration-approved manufacturer's label

SUMMARY:
The primary objective of the study was to characterize the difference in prepubescent growth velocity in children 3 to 9 years of age with perennial allergic rhinitis (PAR) treated with triamcinolone acetonide (TAA) nasal spray (NASACORT® AQ 110 μg treatment group) or placebo (NASACORT® AQ placebo group) for 12-months.

The secondary objectives were to compare the following in prepubertal participants treated with TAA nasal spray versus placebo:

* the 24-hour urinary free cortisol levels and the cortisol/creatinine ratio (to measure the Hypothalamic-Pituitary Adrenal [HPA] axis function)
* the rate of treatment-emergent-adverse-events (TEAE)
* global efficacy rated by the investigator and the participant separately
* the rate of use of rescue medication during the study

DETAILED DESCRIPTION:
The study consisted of:

* a 4- to 6-month screening/baseline period
* a 12-month (up to Day 360+/-5 days) double-blind treatment period starting on Day 1
* a 2-month follow-up period (up to Day 420+/-5 days)

ELIGIBILITY:
Participants meeting the following eligibility criteria were enrolled.

Inclusion criteria:

1. Male participants [3 years to <= 9 years + 0 days old] at Visit 1 and no older than [9 years + 120 days] at Visit 3; and, female participants [3 years to <= 8 years + 0 days old] at Visit 1 and no older than [8 years + 120 days] at Visit 3: all sexually prepubertal (ie, Stage 1 of Tanner Classification of sexual maturity) at Visit 1 and Visit 3. A 5-day extension to the age upper bound was permitted under certain circumstances to enable scheduling of Visits 1 and 3
2. At least a one year history of PAR as assessed and documented by the investigator (with or without seasonal allergic rhinitis [SAR])
3. Positive skin test (prick or intradermal) to a perennial allergen that was present in the participant's environment. A skin test was considered positive if the wheal produced by the allergen was equal to or greater than that caused by positive control (histamine) or was at least 3 mm (prick test) or 7 mm (intradermal test) greater than the wheal of negative control (saline). If a skin test could not be performed, the radioallergosorbent test (RAST) would be used as an alternative. Documented historical skin testing or RAST performed during the past year were acceptable
4. Height within the 3rd and 97th percentiles at screening (Visit 1), Visit 2, and at randomization (Visit 3)
5. Symptomatic (daily AM instantaneous total nasal symptom score was >= 4 out of 12) on any 4 out of the last 7 consecutive days immediately prior to and including the morning of Visit 3. Symptom ratings were to be completed with the help of a parent/guardian/caregiver
6. Written informed consent and ability of parent or legal guardian of the participant to give a written informed consent before any study related procedures. Participants 7 years of age and older must have provided a signed assent form
7. Participants had to be toilet-trained

Exclusion criteria:

1. Gross nasal anatomical deformities including large polyposis and marked deviated septum
2. History of or current cataract or glaucoma
3. History of hypersensitivity to the corticosteroids or to any excipient of the investigational product
4. Participant was the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
5. Height, weight, or body mass index (BMI)-for-age below the 3rd or above the 97th percentile at Visits 1, 2, or 3
6. Treatment with systemic corticosteroids (oral, intravenous, intramuscular, or intra-articular) within 3 months prior to Visit 1
7. Treatment with systemic corticosteroids for >2 courses received up to 1 year before Visit 1 was exclusionary. Up to 2 courses of systemic corticosteroids each course not exceeding 14 days up to 1 year before Visit 1 was allowed.
8. Treatment with inhaled, intranasal, or high potency topical corticosteroid exposure within 6 weeks prior to Visit 1. Mild asthma that was well-controlled and without the use of inhaled corticosteroids within 6 weeks before screening (Visit 1).
9. Immunotherapy, except stable (>=1 month) maintenance schedule before Visit 1.
10. Treatment with any substance before Visit 1 that might have affected growth velocity and/or linear growth, such as, but not be limited to methylphenidate hydrochloride, thyroid hormone, growth hormone, anabolic steroids, calcitonin, estrogens, progestins, bisphosphonates, anticonvulsants, or phosphate-binding antacids
11. Treatment with any investigational product or device in the 30 days before Visit 1 or at any time throughout the duration of this trial (Visit 1 through Visit 11).
12. Bone age as assessed by X-ray of the left hand and wrist that was outside +/- 1.5 years of participants chronological age at Visit 2. Right hand and wrist were to be radiographed in the event of bone injury to the left hand or wrist.
13. Unresolved upper respiratory tract infection, sinus infection or nasal candidiasis (i.e., symptomatic or under treatment) within the last 2 weeks before Visit 3.
14. Participants or parent/guardian/caregiver unable to demonstrate correct administration of the investigational product at Visit 1.
15. Concomitant disease other than PAR which could have interfered with the study procedures or outcomes as determined by the investigator.
16. History of hospitalization due to asthma within 1 year before screening (Visit 1).
17. Abnormal 24-hour urinary free cortisol level assessed at screening (Visit 2).

The above information was not intended to contain all considerations relevant to potential participation in a clinical trial.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 299 (Actual)
Dates: Start 2007-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akbar Akbary, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 14 March 2007 (first subject enrolled) and 12 October 2011 (last subject last visit) at 69 active centers located in the US.
Pre-assignment Details: 299 participants were randomized, 298 were treated.
Groups:
- Placebo: 3 to 9 year old participants with PAR administered
  * Placebo (once to demonstrate IP administration in the baseline/screening period)
  * Placebo in the double-blind treatment period
  All participants were provided Children's Claritin® Syrup as a rescue medication
- TAA-AQ: 3 to 9 year old participants with PAR administered
  * Placebo (once to demonstrate IP administration in the baseline/screening period)
  * TAA-AQ in the double-blind treatment period
  All participants were provided Children's Claritin® Syrup as a rescue medication
Period: Overall Study
Arm/Group | Placebo | TAA-AQ
Started | 148 | 151
Completed | 107 | 109
Not Completed | 41 | 42
Not completed — Adverse Event | 3 | 1
Not completed — Protocol Violation | 14 | 12
Not completed — Lost to Follow-up | 5 | 7
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Lack of Efficacy | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Not treated | 0 | 1
Not completed — Excluded medication | 0 | 2
Not completed — Non-compliance | 2 | 5
Not completed — Sponsor decision | 1 | 3
Not completed — Relocation | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TAA-AQ | Total
Number analyzed (Participants) | 148 | 151 | 299
Age Continuous [Mean (Standard Deviation); unit: years] — Age at screening
  years | 6.24 (1.55) | 6.12 (1.62) | 6.18 (1.58)
Age, Customized [Number; unit: participants] — Age group at screening.
  participants
    <=3 to <6 years | 64 | 65 | 129
    <=6 to <10 years | 84 | 86 | 170
Sex/Gender, Customized [Number; unit: participants]
  Male | 86 | 87 | 173
  Female | 62 | 64 | 126
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/White | 114 | 111 | 225
  Black | 22 | 28 | 50
  Asian/Oriental | 4 | 1 | 5
  American Indian or Alaska Native | 0 | 1 | 1
  Native Hawaiian or other Pacific Island | 0 | 0 | 0
  Other | 8 | 10 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 23 | 33 | 56
  Not Hispanic or Latino | 125 | 118 | 243
Tanner classification at randomization [Number; unit: participants] — Tanner classification distinguishes stages of puberty. Each stage differentiates the extent of breast, genitalia and pubic hair growth. Tanner Stage I represents the preadolescent stage where breast, genitalia and pubic hair growth are of the same size and shape as in early childhood; and in Tanner Stage 5 breasts and genitalia are of adult shape and size, and pubic hair is adult in quantity (mature stage). Stages 2, 3 and 4 are intermediate stages.
  participants
    Stage 1 | 148 | 151 | 299
    Stage 2 | 0 | 0 | 0
    Stage 3 | 0 | 0 | 0
    Stage 4 | 0 | 0 | 0
    Stage 5 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Growth Velocity
Description: Individual participant's growth velocity over double-blind treatment period was calculated using a linear regression of height over time.
  Height was measured on the same wall-mounted Harpenden stadiometer with the participant barefoot and in light clothing.
Time Frame: Day 1 to end of treatment (Day 360)
Population: The modified intent-to-treat (mITT) population included all intent-to-treat participants who had at least 3 postrandomization visits with recorded height measurements during the double-blind treatment period, excluding those from Good Clinical Practice (GCP) noncompliant sites.
Measure: Least Squares Mean (Standard Error); unit: cm/year
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 133 | 134
cm/year | 6.09 (0.122) | 5.65 (0.122)
Statistical Analysis 1: Comparison: Placebo vs TAA-AQ; Test type: Superiority or Other; p = 0.0096, ANCOVA; The treatment arm, age group (at Visit 1) and sex were fixed effects, and baseline growth velocity was a covariate in the ANCOVA model; Difference (LS Mean) = -0.45, 95% CI 2-sided [-0.78 to -0.11]

2. Secondary Outcome: Change From Baseline in Instantaneous Total Nasal Symptom Score (TNSS)
Description: PAR symptoms - nasal stuffiness, nasal discharge, sneezing, and nasal itching were scored upon arising in the morning according to the following 4-point scale:
  * 0 = symptom absent
  * 1 = mild (present but not annoying to self)
  * 2 = moderate (annoying to self but not interfering with sleep or daily living)
  * 3 = severe (interfered with daily living and/or sleep)
  TNSS was the sum of the individual symptom scores (ranging 0-3), and TNSS ranged from 0 (best outcome) to 12 (worst outcome). A negative value for change represents an improvement in symptoms.
Time Frame: For 7 days prior to randomization (Baseline) and everyday for 7 days prior to Day 360 (end of treatment)
Population: mITT population with scores available for TNSS: All randomized and treated participants with at least 3 post-randomization height measurements during the double-blind treatment period with scores available for TNSS, excluding those from GCP noncompliant sites.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 102 | 104
score on a scale | -2.68 (0.26) | -2.80 (0.25)
Statistical Analysis 1: Comparison: Placebo vs TAA-AQ; Test type: Superiority or Other; p = 0.7341, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.83 to 0.58] — The treatment arm, sex and age group were fixed effects, and baseline value was a covariate in the ANCOVA model

3. Secondary Outcome: Change From Baseline in Four Individual Nasal Symptom Scores at the End of Treatment
Description: PAR symptoms - nasal stuffiness, nasal discharge, sneezing, and nasal itching were scored upon arising in the morning according to the following 4-point scale:
  * 0 = symptom absent
  * 1 = mild (present but not annoying to self)
  * 2 = moderate (annoying to self but not interfering with sleep or daily living)
  * 3 = severe (interfered with daily living and/or sleep)
  Individual symptom scores ranged from 0 (best outcome) to 3 (worst outcome). A negative value for change represents an improvement in symptoms.
Time Frame: For 7 days prior to randomization (Baseline) and everyday for 7 days prior to Day 360 (end of treatment)
Population: mITT population with available nasal symptom scores: All randomized and treated participants with at least 3 post-randomization height measurements during the double-blind treatment period with available nasal symptom scores, excluding those from GCP noncompliant sites.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 133 | 134
score on a scale
  Change in Nasal stuffiness (N=101, N=104) | -0.68 (0.08) | -0.83 (0.08)
  Change in Nasal discharge (N=102, N=103) | -0.67 (0.07) | -0.71 (0.07)
  Change in Sneezing (N=102, N=103) | -0.64 (0.07) | -0.55 (0.07)
  Change in Nasal Itching (N=101, N=104) | -0.69 (0.08) | -0.71 (0.08)
Statistical Analysis 1: Comparison: Placebo vs TAA-AQ; Change in nasal stuffiness; Test type: Superiority or Other; p = 0.1963, ANCOVA; LS Mean Differerence = -0.15, 95% CI 2-sided [-0.37 to 0.08] — The treatment arm, sex and age group were fixed effects, and baseline value was a covariate in the ANCOVA model
Statistical Analysis 2: Comparison: Placebo vs TAA-AQ; Change in Nasal Discharge; Test type: Superiority or Other; p = 0.7193, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.24 to 0.17] — The treatment arm, sex and age group were fixed effects, and baseline value was a covariate in the ANCOVA model
Statistical Analysis 3: Comparison: Placebo vs TAA-AQ; Change in Sneezing; Test type: Superiority or Other; p = 0.4020, ANCOVA; LS Mean Difference = 0.09, 95% CI 2-sided [-0.12 to 0.29] — The treatment arm, sex and age group were fixed effects, and baseline value was a covariate in the ANCOVA model
Statistical Analysis 4: Comparison: Placebo vs TAA-AQ; Change in Nasal Itching; Test type: Superiority or Other; p = 0.8854, ANCOVA; LS mean Difference = -0.02, 95% CI 2-sided [-0.23 to 0.20] — The treatment arm, sex and age group were fixed effects, and baseline value was a covariate in the ANCOVA model

4. Secondary Outcome: Global Efficacy as Assessed by the Participant (With the Help of a Parent/Guardian/Caregiver) During and at the End of the Double-blind Treatment Period
Description: Global efficacy was assessed by the participant (with the help of a parent/guardian/caregiver) using the following scale:
  * 0 = no relief (symptoms unchanged or worse than before)
  * 1 = slight relief (symptoms were present and only minimally improved)
  * 2 = moderate relief (symptoms were present and could have been troublesome but were noticeably improved)
  * 3 = marked relief (symptoms were greatly improved and although present were scarcely troublesome)
  * 4 = complete relief (virtually no symptom present)
Time Frame: Day 120, Day 240 and Day 360
Population: mITT population: All randomized and treated participants with at least 3 post-randomization height measurements during the double-blind treatment period, excluding those from GCP noncompliant sites.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 133 | 134
score on a scale
  Day 120 (N=127, N=131) | 1.87 (1.10) | 2.09 (1.00)
  Day 240 (N=115, N=116) | 1.97 (1.04) | 2.16 (1.03)
  Day 360 (N=125, N=125) | 1.86 (1.08) | 2.18 (1.19)
Statistical Analysis 1: Comparison: Placebo vs TAA-AQ; Statistical Analysis for Day 120; Test type: Superiority or Other; p = 0.0951, Mixed model for repeated measures; The treatment arm, assessment visit, their interaction, sex and age group were fixed effects, and assessment visit was a repeated factor
Statistical Analysis 2: Comparison: Placebo vs TAA-AQ; Statistical analysis for Day 240; Test type: Superiority or Other; p = 0.1247, Mixed model for repeated measures; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAA-AQ; Statistical analysis for Day 360; Test type: Superiority or Other; p = 0.0207, Mixed model for repeated measures; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Global Efficacy as Assessed by the Investigator During and at the End of the Double-blind Treatment Period
Description: Global efficacy was assessed by the investigator using the following scale:
  * 0 = no relief (symptoms unchanged or worse than before)
  * 1 = slight relief (symptoms were present and only minimally improved)
  * 2 = moderate relief (symptoms were present and could have been troublesome but were noticeably improved)
  * 3 = marked relief (symptoms were greatly improved and although present were scarcely troublesome)
  * 4 = complete relief (virtually no symptom present)
Time Frame: Day 120, Day 240 and Day 360
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 133 | 134
score on a scale
  Day 120 (N=128, N=130) | 1.89 (1.11) | 2.04 (1.04)
  Day 240 (N=115, N=136) | 2.11 (1.07) | 2.21 (1.08)
  Day 360 (N=125, N=125) | 1.80 (0.98) | 2.14 (1.16)
Statistical Analysis 1: Comparison: Placebo vs TAA-AQ; Statistical Analysis for Day 120; Test type: Superiority or Other; p = 0.2445, Mixed model for repeated measures; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TAA-AQ; Statistical Analysis for Day 240; Test type: Superiority or Other; p = 0.4488, Mixed model for repeated measures; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAA-AQ; Statistical Analysis for Day 360; Test type: Superiority or Other; p = 0.0142, Mixed model for repeated measures — The treatment arm, assessment visit, their interaction, sex and age group were fixed effects, and assessment visit was a repeated factor

6. Secondary Outcome: Percentage of Participants Who Used the Rescue Medication During the Double-blind Phase of the Study
Description: Children's Claritin® syrup was provided as a rescue medication to control allergic rhinitis (AR) symptoms and could be used throughout the study on an as needed basis. Use of rescue medication was to be documented in the participant's diary.
  The percentage of participants who used the rescue medication during each of the study periods is reported.
Time Frame: Baseline (4-6 months before Day 1), double-blind treatment period (Day 1 to Day 360) and follow-up (Day 361 to Day 420)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 133 | 134
percentage of participants | 81.2 | 90.3

7. Secondary Outcome: Percentage of Days Participants Used the Rescue Medication During the Double-blind Treatment Phase of the Study
Description: Children's Claritin® syrup was provided as a rescue medication to control allergic rhinitis (AR) symptoms and could be used throughout the study on an as needed basis. Use of rescue medication was to be documented in the participant's diary.
  The percentage of days that participants used the rescue medication during the double-blind treatment phase of the study.
Time Frame: double-blind treatment period (Day 1 to Day 360)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 133 | 134
percentage of days | 20.39 (28.02) | 15.69 (21.53)

8. Secondary Outcome: 24 Hour Urinary Free Cortisol Levels
Description: Urine cortisol levels was determined at screening, at the end of treatment, and at follow-up visit using routine laboratory testing. The normal range for urinary free cortisol for 3- to 9-year-olds was considered to be [1.4 - 21 μg/24 hours].
Time Frame: Baseline (2 to 6 weeks before Day 1), end of treatment (Day 360), and at follow-up (Day 420)
Population: All randomized and treated participants, excluding those from GCP noncompliant sites.
Measure: Mean (Standard Deviation); unit: μg/24 hours
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 147 | 146
μg/24 hours
  at baseline (N=146, N=141) | 7.44 (4.23) | 7.44 (4.04)
  at end of treatment (EOT) (N=114, N=118) | 7.05 (5.33) | 7.42 (5.93)
  at follow-up (N=96, N=97) | 7.85 (5.65) | 7.00 (5.28)

9. Secondary Outcome: 24 Hour Cortisol/Creatinine Ratio
Description: Urine cortisol and creatinine levels were determined at screening, at the end of treatment, and at follow-up visit using routine laboratory testing. The normal range for urinary free cortisol for 3- to 9-year-olds was considered to be [1.4 - 21 μg/24 hours]. No normal range is available for cortisol/creatinine ratio.
Time Frame: Baseline (2 to 6 weeks before Day 1), end of treatment (Day 360), and at follow-up (Day 420)
Population: All randomized and treated participants, excluding those from GCP noncompliant sites.
Measure: Mean (Standard Deviation); unit: μg/g Creatinine
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 147 | 146
μg/g Creatinine
  at baseline (N=145, N=141) | 18.94 (9.64) | 19.44 (10.62)
  at end of treatment (N=114, N=118) | 15.47 (12.60) | 15.86 (10.77)
  at follow-up (N=96, N=97) | 17.01 (12.63) | 15.10 (9.54)

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: Adverse events that developed, worsened, or became serious during the double-blind treatment period or within 7 days after the last dose of double-blind investigational product (IP) are defined as TEAEs.
  A serious adverse event (SAE) was defined as any untoward medical occurrence that at any dose:
  * Resulted in death
  * Was life-threatening
  * Required inpatient hospitalization or prolongation of existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * Was a congenital anomaly/birth defect
  * Was a medically important event
Time Frame: From Day 1 to 7 days following end of treatment (Day 360)
Population: All randomized and treated participants, excluding those from GCP noncompliant sites.
Measure: Number; unit: participants
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 147 | 146
participants
  with any TEAE | 113 | 117
  with any treatment emergent SAE | 0 | 2
  with any TEAE leading to permanent discontinuation | 3 | 1
  with any TEAE leading to death | 0 | 0
  with investigational product (IP) overdose TEAE | 0 | 0

ADVERSE EVENTS:
Time Frame: From treatment initiation to 7 days after the last dose of double-blind treatment (double blind treatment period)
Description: Adverse events that developed, worsened, or became serious during the double-blind treatment period or within 7 days after the last dose of double-blind period, i.e. Treatment-emergent adverse events.
Arm/Group | Placebo | TAA-AQ
Serious Adverse Events (participants affected / at risk) | 0/147 | 2/146
Other Adverse Events (participants affected / at risk) | 98/147 | 109/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=147) | TAA-AQ (N=146)
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=147) | TAA-AQ (N=146)
Nasopharyngitis (Infections and infestations) | 18 | 28
Upper respiratory tract infection (Infections and infestations) | 19 | 25
Pharyngitis streptococcal (Infections and infestations) | 10 | 12
Sinusitis (Infections and infestations) | 11 | 12
Influenza (Infections and infestations) | 3 | 10
Viral infection (Infections and infestations) | 3 | 9
Viral upper respiratory tract infection (Infections and infestations) | 9 | 9
Gastroenteritis viral (Infections and infestations) | 6 | 8
Otitis media (Infections and infestations) | 8 | 4
Headache (Nervous system disorders) | 31 | 34
Ear pain (Ear and labyrinth disorders) | 14 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 29
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 16
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Vomiting (Gastrointestinal disorders) | 8 | 19
Abdominal pain upper (Gastrointestinal disorders) | 15 | 16
Rash (Skin and subcutaneous tissue disorders) | 4 | 10
Pyrexia (General disorders) | 37 | 31

LIMITATIONS AND CAVEATS:
Two study sites with significant GCP noncompliance were reported to the U.S. Food and Drug Administration (FDA) by the Sponsor. A total of 5 treated participants (1 placebo and 4 TAA-AQ) from these 2 study sites were excluded from the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can independently publish study results from his site after the primary publication by the steering committee, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication derived from the study for review and comment at least 45 days (20 days for abstracts) in advance of any submission, and delay publication till the approval of the publication is given in writing by the Sponsor (not to exceed ninety days).